CLINICAL TRIAL: NCT03218410
Title: Surgical Pulmonary Embolectomy Versus Catheter-directed Thrombolysis in the Treatment of Pulmonary Embolism: A Randomized Phase II Non-inferiority Study
Brief Title: Surgical Pulmonary Embolectomy Versus Catheter-directed Thrombolysis in the Treatment of Pulmonary Embolism: A Non-inferiority Study
Acronym: Lungembolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other); Schweizerische Herzstiftung (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 183/15
Record Dates: First submitted 2017-07-13; First posted 2017-07-14 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Acute Pulmonary Embolism (PE)
Keywords: surgical embolectomy; catheter-directed therapy

STUDY DESIGN:
Intervention Model Description: Monocentric, randomized, open-label, controlled, clinical, non-inferiority trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgical pulmonary embolectomy (Active Comparator)
  Interventions: Procedure: surgical pulmonary embolectomy
- catheter-directed thrombolysis (Active Comparator)
  Interventions: Combination Product: catheter-directed thrombolysis

INTERVENTIONS:
Procedure: surgical pulmonary embolectomy
  Arms: surgical pulmonary embolectomy
Combination Product: catheter-directed thrombolysis
  Arms: catheter-directed thrombolysis

SUMMARY:
Acute pulmonary embolism (PE) is a serious and potentially lethal condition. The clinical spectrum of PE spans from asymptomatic PE to patients with severe hemodynamic compromise. The main determinant of outcome is right ventricular dysfunction caused by the abrupt rise in pulmonary vascular resistance. Patients with hemodynamic compromise are at highest risk of mortality (>15%). Hemodynamic stable patients with imaging and biomarker evidence of right ventricular (RV)- dysfunction are at intermediate-high risk of mortality (3-15%). According to the European Society of Cardiology (ESC) guidelines reperfusion therapy options for patients at high risk and at intermediate-high risk include systemic thrombolysis, catheter-directed therapy or surgical embolectomy.

The University Hospital of Bern is the only tertiary care hospital in Switzerland that has established an interdisciplinary pulmonary embolism response team (PERT since 2010) and has gained expertise in both catheter-directed thrombolysis and surgical embolectomy. Since the introduction of PERT, systemic thrombolysis was no longer performed in Bern due to the high risk of intracranial hemorrhage. Favorable clinical outcomes of the patients managed in Bern have been published for both catheter-directed therapy and surgical embolectomy.

To date, no study has ever compared catheter-directed thrombolysis versus surgical pulmonary embolectomy in the treatment of high and intermediate-high risk PE patients.

DETAILED DESCRIPTION:
Background and Study Rationale:

Acute pulmonary embolism (PE) is a serious and potentially lethal condition. The clinical spectrum of PE spans from asymptomatic PE to patients with severe hemodynamic compromise. The main determinant of outcome is right ventricular dysfunction caused by the abrupt rise in pulmonary vascular resistance. Patients with hemodynamic compromise are at highest risk of mortality (>15%). Hemodynamic stable patients with imaging and biomarker evidence of right ventricular (RV)- dysfunction are at intermediate-high risk of mortality (3-15%). According to the European Society of Cardiology (ESC) guidelines reperfusion therapy options for patients at high risk and at intermediate-high risk include systemic thrombolysis, catheter-directed therapy or surgical embolectomy.

The University Hospital of Bern is the only tertiary care hospital in Switzerland that has established an interdisciplinary pulmonary embolism response team (PERT since 2010) and has gained expertise in both catheter-directed thrombolysis and surgical embolectomy. Since the introduction of PERT, systemic thrombolysis was no longer performed in Bern due to the high risk of intracranial hemorrhage. Favorable clinical outcomes of the patients managed in Bern have been published for both catheter-directed therapy and surgical embolectomy.

To date, no study has ever compared catheter-directed thrombolysis versus surgical pulmonary embolectomy in the treatment of high and intermediate-high risk PE patients.

Primary Objective:

Non-inferiority of catheter-directed thrombolysis to surgical pulmonary embolectomy regarding efficacy in reversal of RV dilatation in high and intermediate -high risk patients with acute pulmonary embolism.

Number of Patients:

60 patients (30 with surgical pulmonary embolectomy and 30 with catheter-directed thrombolysis therapy) Number of Centers: 1

Study Patient Treatment:

All patients will receive standard anticoagulant therapy. In a 1:1 fashion, patients will be randomized to undergo catheter-directed thrombolysis or surgical pulmonary embolectomy. Stratification will be performed by the presence of high-risk pulmonary embolism.

Trial Duration: 24 months Start Date: October 2015 Stop Date: June 2017 Publication: 2017 Standard Therapy Anticoagulation is the main therapy for acute PE once the diagnosis is established. The main objectives of anticoagulant therapy in the initial treatment are to prevent thrombus extension and secondary recurrence of venous thromboembolism. Current guidelines recommend an initial treatment for at least 5 days with either subcutaneous low-molecular-weight heparin (LMWH), intravenous or subcutaneous unfractioned heparin, or subcutaneous fondaparinux as well as the initiation of oral vitamin-K antagonists at the same time. 6 In addition to anticoagulation, the recent European Society of Cardiology (ESC) guidelines recommend systemic thrombolysis in PE patients at high risk of death (Grade 1B) and should be considered in patients at intermediate-high risk of death.6 However, recent evidence shows that hemodynamic decompensation is prevented in patients with intermediate-high risk PE, but the incidence of major bleeding complications (20%) and intracranial hemorrhage (up to 3%) increased significantly.8 Therefore systemic fibrinolytic therapy is withheld in the majority of cases mainly due to the fear of life-threatening bleeding complications including intracranial hemorrhage. 4 Due to the high risk of intracranial bleeding complications, systemic thrombolysis therapy is no longer performed at the Inselspital Bern.

Given that high and intermediate-high risk PE patients require special attention, a standardized procedure is provided to these patients by an established pulmonary embolism response team (PERT) at the Inselspital in Bern. The pulmonary embolism response team consists of an angiologist, a cardiologist, an emergency physician, and a cardiac surgeon available 24 hours a day, and 7 days a week. Each patient is evaluated whether he/she is best treated by anticoagulation only or additional catheter-directed thrombolysis or surgical pulmonary embolectomy is indicated. Hereby, an already established standardized clinical algorithm is used to guide treatment procedures depending on the individual risk setting (Appendix 5).

It should be emphasized, that this clinical pathway in Bern is only possible due to the fact, that there is an experienced interdisciplinary and standardized approach to patients with pulmonary embolism. Pulmonary embolism response teams (PERT) are established in several academic hospitals in the United States of America, including the Brigham and Women's Hospital and the Massachusetts General Hospital, both in Boston, Harvard Medical School. The University Hospital Bern has established the first interdisciplinary PERT in Europe in 2010 and remains the only European academic hospital offering both surgical embolectomy and catheter therapy on a 24 basis to patients with acute pulmonary embolism at increased risk of death. The Cardiovascular Center of the University Hospital Bern belongs to one of the few hospitals worldwide that has clinical experience in both surgical embolectomy and catheter therapy. Excellent clinical results were published for both techniques. Therefore, the University Hospital Bern has the unique opportunity to perform a randomized controlled clinical trial and compare both techniques. A large multicenter trial powered for a mortality analysis would be ideal to investigate the efficacy and safety of both techniques. A clinical trial designed for non-inferiority would require more than 1000 patients enrolled from over 50 centers. However, due to the fact that PERTs are not yet established in Europe, we intend to perform a single center study in Bern using surrogate endpoints, i.e. reversal of right heart failure and reduction in thrombus load. The study will not be powered for clinical endpoints but will assess secondary endpoints, including mortality, bleeding complications, exercise performance, and quality of life up to 12 months after the revascularization procedure.

Revascularization Strategies The main objective of early revascularization strategies in patients with PE is to reduce the thrombus load in pulmonary arteries, thereby reversing right ventricular dysfunction improving symptoms and survival.9 Reperfusion strategies encompass catheter-directed thrombolysis and surgical embolectomy and should be considered in selected high and intermediate-high-risk patients with PE.

According to current guidelines of the European Society of Cardiology (ESC) published in 20146 catheter-directed treatment (Grade 2aC) or surgical embolectomy (Grade 1C) should be considered in all patients with PE at high risk, in whom systemic thrombolytic therapy is contraindicated or has failed. Also, catheter-directed treatment (Grade 2bB) or surgical embolectomy (Grade 2bC) may be considered in intermediate-high-risk patients with PE. However, it remains unclear, which reperfusion strategy is most appropriate for high and intermediate-high-risk patients with PE.

Catheter-directed Thrombolysis Given, that anticoagulation alone has little effect on improvement of RV performance in the early phase, catheter-directed thrombolysis appears to be effective for early RV recovery.10 There are two main approaches for catheter-directed thrombolysis, i.e., conventional catheter-directed thrombolysis and pharmacomechanical thrombolysis.

Conventional catheter-directed thrombolysis:

Thrombolytic agents, for example, recombinant tissue plasminogen activator (rtPA) at a dose of 1-2mg per hour for up to 24 hours, are infused through side-hole catheters which are placed at the side of the thrombotic occlusion in the pulmonary arteries.

Pharmacomechanical thrombolysis:

Pharmacomechanical thrombolysis refers to catheter-directed thrombolysis combined with a mechanical catheter technique. In addition to the thrombectomy mode, the AngioJet® system (Boston Scientific, USA) enables a high-pressure intraclot injection of thrombolytic agents (PowerPulse® technique). Ultrasound-assisted thrombolysis is another type of pharmacomechanical thrombolysis which aims to accelerate thrombolysis success. It consists of a thrombolysis catheter with a microsonic core wire that uses high-frequency low-power ultrasound waves (EKOS Corporation; Bothell, WA, USA).

In a randomized, controlled clinical trial of 59 intermediate-risk patients ultrasound assisted catheter-directed- thrombolysis significantly reduced RV-LV ratio after 24 hours compared to heparin alone without an increase in bleeding rates.11 In the present trial, pharmacomechanical thrombolysis will be used in the catheter therapy group.

Surgical Pulmonary Embolectomy Historically and according to current guidelines, surgical embolectomy (SE) is reserved for patients in whom thrombolysis was contraindicated or had failed. Therefore the majority of SE were performed in critically ill patients, resulting in high mortality rates.12 Recent publications including our own experience reported reduced mortality rates even in patients with cardiac arrest and preoperative cardiopulmonary resuscitation13. Many authors question the restrictive role of SE compared to systemic thrombolytic therapy and advocate SE in hemodynamically stable patients with signs of RV Dysfunction and high clot burden in the central pulmonary artery.

Surgical embolectomy (SE) is performed though a median sternotomy using mild hypothermic or normothermic cardiopulmonary bypass (CPB). The main pulmonary artery is opened with a longitudinal incision, which can be extended into the right and left pulmonary artery branches. The thrombotic material is extracted using a special forceps and by assisting suction. To ensure complete clot removal the right and left pulmonary artery branches a flexible surgical angioscope can be used to inspect the segmental arteries. Massage of the lungs is not performed to avoid additional damage to the lung parenchyma. The right atrium and ventricle are routinely explored, all clot material is carefully removed and a patent foramen ovale if present is closed with a 4-0 running suture. The pulmonary arteriotomy is closed with a running suture, and the patient is weaned from CBP after declamping of the aorta. The patient is transferred to the intensive care unit and is treated with intravenous unfractioned heparin (initial dosage of 1000Ul/24h, the goal is to achieve an activated partial thromboplastin-time ratio of at least twice the control value) starting six hours after surgery. All patients receive in the follow-up period oral anticoagulation with warfarin (starting on postoperative day one) with an International Normalized Ratio (INR) target of 2.5± 0.5 for at least 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Acute symptomatic PE with thrombus located in the pulmonary main trunk or the left and/or right main pulmonary artery
2. High-risk PE defined as PE with sustained systemic arterial hypotension (systolic pressure <90mmHg), cardiogenic shock, or the ongoing need for catecholamine therapy

   OR

   Intermediate-high risk PE: Imaging evidence of RV-Dilatation (right-to-left ventricular diameter ratio >1.0 on echocardiography or chest computed tomography) and biomarker evidence of RV dysfunction (positive Troponin T or I Test).
3. The eligibility for both procedures must be established by the PERT team
4. Signed Informed consent (by subject or legal representative) -

Exclusion Criteria:

1. Age less than 18 years or greater than 80 years.
2. Symptom duration > 14 days suggesting acute-on-chronic pulmonary embolism.
3. Known chronic thromboembolic pulmonary hypertension (CTEPH)
4. Suspected chronic thromboembolic pulmonary hypertension (CTEPH) including RV hypertrophy (RV free wall >5 mm on echocardiography), severe pulmonary hypertension (systolic pulmonary artery pressure > 80 mmHg on echocardiography), or CT findings suggestive of CTEPH including intraluminal webs, bands, strictures, or eccentric filling defects adjacent to the wall of the pulmonary arteries
5. Decompensated cardiogenic shock defined as recent (<48 hours) cardiopulmonary resuscitation therapy or worsening hemodynamic status despite extended fluid and catecholamine support
6. Inability to tolerate catheter procedure or surgical embolectomy due to severe comorbidities.
7. Allergy, hypersensitivity, or thrombocytopenia from heparin, r-tPA, or iodinated contrast, except for mild-moderate contrast allergies for which steroid pre-medication can be used.
8. Known significant bleeding risk, or known coagulation disorder (including vitamin K antagonists with INR > 2.0 and platelet count < 100 000/mm3)
9. Severe renal impairment (estimated GFR < 30 ml/min).
10. Active bleeding: recent (< 3 months) GI bleeding, severe liver dysfunction, bleeding diathesis.
11. Recent (< 3 months) internal eye surgery or hemorrhagic retinopathy; recent (< 10 days) major surgery, cataract surgery, trauma, CPR, obstetrical delivery, or other invasive procedure.
12. History of stroke or intracranial/intraspinal bleed, tumor, vascular malformation, aneurysm.
13. Severe hypertension on repeated readings (systolic > 180 mmHg or diastolic > 105 mmHg).
14. Pregnant, lactation or parturition within the previous 30 days (positive pregnancy test in women of childbearing age)
15. Recent (< 1 month) systemic thrombolysis.
16. Life expectancy < 6 months or chronic non-ambulatory status.
17. Participating in any other investigational drug or device study or previous enrollment in this study
18. Inability to comply with study assessments (e.g. due to cognitive impairment or geographic distance).
19. Any other condition that the investigator feels would place the patient at increased risk if the investigational therapy is initiated.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Difference in RV/LV ratio by contrast-enhanced chest computed tomography | 48-72 hours after surgical embolectomy or catheter therapy

SECONDARY OUTCOMES:
Difference in pulmonary occlusion score by contrast-enhanced chest computed tomography | 48-72 hours after surgical embolectomy or catheter therapy

CONTACTS AND LOCATIONS:
Overall Officials: Lars Englberger, Prof., Principal Investigator — University of Bern
Locations (1):
- University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Laporte S, Mismetti P, Decousus H, Uresandi F, Otero R, Lobo JL, Monreal M; RIETE Investigators. Clinical predictors for fatal pulmonary embolism in 15,520 patients with venous thromboembolism: findings from the Registro Informatizado de la Enfermedad TromboEmbolica venosa (RIETE) Registry. Circulation. 2008 Apr 1;117(13):1711-6. doi: 10.1161/CIRCULATIONAHA.107.726232. Epub 2008 Mar 17. PMID 18347212
- [Result] Silverstein MD, Heit JA, Mohr DN, Petterson TM, O'Fallon WM, Melton LJ 3rd. Trends in the incidence of deep vein thrombosis and pulmonary embolism: a 25-year population-based study. Arch Intern Med. 1998 Mar 23;158(6):585-93. doi: 10.1001/archinte.158.6.585. PMID 9521222
- [Result] Cohen AT, Agnelli G, Anderson FA, Arcelus JI, Bergqvist D, Brecht JG, Greer IA, Heit JA, Hutchinson JL, Kakkar AK, Mottier D, Oger E, Samama MM, Spannagl M; VTE Impact Assessment Group in Europe (VITAE). Venous thromboembolism (VTE) in Europe. The number of VTE events and associated morbidity and mortality. Thromb Haemost. 2007 Oct;98(4):756-64. doi: 10.1160/TH07-03-0212. PMID 17938798
- [Result] Kucher N, Rossi E, De Rosa M, Goldhaber SZ. Massive pulmonary embolism. Circulation. 2006 Jan 31;113(4):577-82. doi: 10.1161/CIRCULATIONAHA.105.592592. Epub 2006 Jan 23. PMID 16432055